CLINICAL TRIAL: NCT04116021
Title: The Analgesic Efficacy of the Pectoral Nerves Block Versus Local Anesthetic Infiltration After Mastectomy: a Randomized, Controlled, Double Blinded Trial
Brief Title: The Analgesic Efficacy of the Pectoral Nerves Block Versus Local Anesthetic Infiltration After Mastectomy
Acronym: PECS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hôpital du Valais (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PECS 2019
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers and outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS block (Active Comparator): Ultrasound-guided pectoral nerve block with bupivacaine 0.5 % 30 mL before surgical incision
  Interventions: Other: PECS block
- Wound infiltration (Active Comparator): Wound infiltration with bupivacaine 0.5 % 30 mL at the end of surgery
  Interventions: Other: Local infiltration

INTERVENTIONS:
Other: PECS block — Ultrasound-guided PECS block before surgical incision with 30 mL bupivacaine 0.5 %
  Arms: PECS block
Other: Local infiltration — Wound infiltration at the end of surgery with with 30 mL bupivacaine 0.5 %
  Arms: Wound infiltration

SUMMARY:
This trial will include patients undergoing radical mastectomy under general anesthesia. One group of patients will receive a pectoral nerve block, done by the anesthetist under ultrasound guidance at the beginning of the invervention. The other group will receive the a wound infiltration at the end of the intervention, done by the surgeon. Investigators will compare acute pain-related outcomes and chronic pain at 3 and 6 months postoperatively.

DETAILED DESCRIPTION:
Mastectomies are associated with moderate to severe postoperative pain. In addition to general anesthesia, different methods of locoregional anesthesia exist to treat postoperative pain, amongst others a pectoral nerve block. This block consists in injecting local anesthetic between the muscles of the thoracic wall and is done under ultrasound guidance. Over the last few years, the pectoral nerves block has become a recognized option for the treatment of acute post-mastectomy pain and it is routinely performed in addition to general anesthesia.

Data indicates that pectoral nerve blocks are effective for the treatment of postoperative pain during the first 24 hours after mastectomy, when compared to no block. However, the analgesic efficacy of a pectoral nerve block has never systematically compared to that of wound infiltration with local anesthetics, done by the surgeon at the end of the intervention. Such an infiltration is also currently employed.

In our study randomize patients undergoing mastectomy under general anesthesia will be randomized to receive either an ultrasound-guided pectoral nerve block with 30 mL of local anesthetic (group PECS) or a wound infiltration with 30 mL of local anesthetic (group infiltration).

Investigators will assess different pain-related outcomes over the first 24 postoperative hours, together with potential block-related side effects and patient satisfaction. Chronic postoperative pain at 3 and 6 months postoperatively will also be assessed.

Both patients and outcome assessors will be blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral mastectomy
* American Society of Anesthesiology Physical Status I-III
* Age ≥ 18

Exclusion Criteria:

* Contraindications to regional anesthesia, such as infection at the surgical site
* Pregnancy
* History of alcohol or drug dependence/abuse
* History of long term opioid intake
* Chronic pain disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | first 24 postoperative hours
  Cumulative intravenous morphine consumption (mg)

SECONDARY OUTCOMES:
Pain score at rest at 2 hours postoperatively | 2 hours postoperatively
  Numeric rating scale from 0 = no pain to 10 = worst imaginable pain
Pain score at rest at 12 hours postoperatively | 12 hours postoperatively
  Numeric rating scale from 0 = no pain to 10 = worst imaginable pain
Pain score at rest at 24 hours postoperatively | 24 hours postoperatively
  Numeric rating scale from 0 = no pain to 10 = worst imaginable pain
Pain score on movement at 2 hours postoperatively | 2 hours postoperatively
  Numeric rating scale from 0 = no pain to 10 = worst imaginable pain
Pain score on movement at 12 hours postoperatively | 12 hours postoperatively
  Numeric rating scale from 0 = no pain to 10 = worst imaginable pain
Pain score on movement at 24 hours postoperatively | 24 hours postoperatively
  Numeric rating scale from 0 = no pain to 10 = worst imaginable pain
Time to first analgesic request | 24 hours postoperatively
  Time between end of surgery and first analgesic request by patient, in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sina Grape, Principal Investigator — Hopital du Valais

IPD SHARING:
Plan to Share IPD: No